CLINICAL TRIAL: NCT06319924
Title: Fixed Low-dose Simethicone Combined With Macrogol 4000 (PEG) Reduces Colon Bubble Formation in Colonoscopy: Phase 4 Prospective Multicenter Real Life Study
Brief Title: Fixed Low-dose Simethicone Combined With Macrogol 4000 (PEG) Reduces Colon Bubble Formation in Colonoscopy
Acronym: XIMEPEG-RL
Status: Completed | Type: Observational
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Sponsor
Other Study IDs: XIMEPEG-RL
Record Dates: First submitted 2024-02-28; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer; Colonoscopy; Bowel Preparation Solution
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Polyethylene Glycols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Simethicone combined with Macrogol 4000 (PEG) — bowel preparation product for colonoscopy as part of CRC screening

SUMMARY:
Several randomised studies have shown that the addition of low-dose Simethicone to the bowel preparation was sufficient to reduce the presence of bubbles during colonoscopy. The aim of this study was to evaluate the efficacy and safety of a bowel preparation containing low-dose Simethicone on bubble formation.

Patients and Methods This prospective, real-life, phase 4 study was conducted from February 2020 to May 2021, in five private endoscopy centres, among adult patients undergoing a colonoscopy. Clinical, endoscopic and histological parameters were collected on e-CRF. The primary endpoint was the measurement of bubble formation in the various colon segments.

ELIGIBILITY:
Inclusion Criteria:

patients :

* scheduled for colonoscopy as part of CRC screening, using the bowel preparation with fixed low-dose of simethicone combined with Macrogol 4000 (PEG)
* aged 50-75 years,
* with no family history of CRC or personal history of colon polyps but with a positive Faecal Immunochemical Test (FIT), with a family history of CRC or personal history of colon polyps,
* requiring surveillance colonoscopy after 5 years if diagnosed with one or two tubular adenomas <10 mm in diameter (low-risk group) or after 3 years if diagnosed with at least 3 adenomas or any adenoma at least 10 mm in diameter or with high-grade dysplasia, according to French recommendations during the study inclusion period.

Exclusion Criteria:

-

Ages: 50 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients, scheduled for colonoscopy as part of CRC screening, were prospectively included according to the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 601 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Assess the quality of the bowel preparation assessed by Bubble scale | During procedure
Assess the quality of the bowel preparation assessed by Boston Bowel Preparation Scale (BBPS) | During procedure

SECONDARY OUTCOMES:
Colonoscope removal time | immediately post procedure
  time spent by the endoscopist searching for polyps and adenomas (mn)
The frequency of adverse events (AEs) | within 10 minutes post procedure
  including nausea, vomiting, abdominal bloating - and their severity,
volume of bowel preparation ingested | immediately post procedure
  in ml
Caecal intubation rate | immediately post procedure.
  successful Caecal intubation

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Clinique des Cèdres, Ramsay Santé,, Cornebarrieu
  - Polyclinique Louis Pasteur,, Essey-lès-Nancy
  - Saint Joseph Hospital, Marseille
  - 5. Clinique Ambroise Paré, Toulouse
  - Pole Santé des Haberges, Vesoul

IPD SHARING:
Plan to Share IPD: No